CLINICAL TRIAL: NCT03541018
Title: Which Repositional Maneuver is the Most Successful When Treating Lateral and Posterior Benign Paroxysmal Positional Vertigo With the TRV Repositional Chair?
Brief Title: Different Treatments With the TRV Reposition Chair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Dan Dupont Hougaard, MD, Assistant Professor, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VEST01
Record Dates: First submitted 2018-05-04; First posted 2018-05-30 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Benign Paroxysmal Positional Vertigo
Keywords: TRV Reposition Chair; Epley Maneuvre
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posterior canalolithiasis (Experimental): Type of repositional maneuvre
  Interventions: Procedure: Type of repositional maneuvre
- Lateral cupulolithiasis (Experimental): Type of repositional maneuvre
  Interventions: Procedure: Type of repositional maneuvre

INTERVENTIONS:
Procedure: Type of repositional maneuvre — Patients randomized to 2 different repositional maneuvres related to the subtypes of BPPV

SUMMARY:
To investigate which treatment option (reposition maneuver) with the TRV chair that is the most effective in patients diagnosed with benign paroxysmal positional vertigo (BPPV). Subtypes of BPPV will be examined after randomization to specific treatments.

DETAILED DESCRIPTION:
Patients diagnosed with BPPV with subtypes of either posterior canalolithiasis or lateral cupulolithiasis will we considered for enrollment. Each subgroup of patients will undergo randomization for a specific treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years of age
* Medical history compatible with BPPV
* Verification of BPPV with either Dix-Hallpike Maneuver or Supine Roll Test.

Exclusion Criteria:

* Former treatment with a repositional Chair
* Not being able to participate or cooperate in the treatment provided by the TRV Repositional Chair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Evaluation by VNG Measurements | 2 years
  Video NystagmoGraphy (VNG) equipment will objectively quantify nystagmus characteristics during diagnostic procedures.
Subjective vertigo | 2 years
  A systematic registration of experienced vertigo during each diagnostic procedure will take place.

SECONDARY OUTCOMES:
Dizziness Handicap Inventory (DHI) questionnaire | 2 years
  Pre-treatment fulfillment of the questionnaire "Dizziness Handicap Inventory" (DHI) will quantify the level of experienced vertigo.

CONTACTS AND LOCATIONS:
Overall Officials: Dan D Hougaard, MD, Principal Investigator — Aalborg University Hospital, Denmark
Locations (1):
- Department of Otolaryngology, Head & Neck Surgery and Audiology, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No